CLINICAL TRIAL: NCT03974152
Title: Effects of Nicotine Salt Aerosol on Cigarette Smokers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID concerns, funding delays led to cancellation of project
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Paul T. Harrell, Associate Professor, Eastern Virginia Medical School
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 19-01-FB-0009; U54DA036105 (NIH); FP00006477_SA007 (Other Grant/Funding Number: Subaward Number)
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Results first posted 2024-02-02 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-02

CONDITIONS: Electronic Cigarette Use
MeSH Terms: conditions — Vaping | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Own brand cigarette first, then ENDS with protonated nicotine, then ENDS with unprotonated nicotine (Experimental): In each of the 3 sessions, participants will be instructed to take one puff of the tobacco product (cigarette or Subox Mini C ENDS with 18 mg nicotine) every 30 seconds for 5 minutes followed by a 2nd blood draw (if staffing allows). Next, participants will be given 90 minutes to use ad lib, i.e., as much as desired.
  Interventions: Other: Subox Mini C with Avail 18 mg nicotine salt (protonated); Other: Subox Mini C with Avail 18 mg nicotine (unprotonated); Other: Own brand cigarette
- ENDS with unprotonated nicotine first, then ENDS with protonated nicotine, then Own brand cigarette (Experimental): In each of the 3 sessions, participants will be instructed to take one puff of the tobacco product (cigarette or Subox Mini C ENDS with 18 mg nicotine) every 30 seconds for 5 minutes followed by a 2nd blood draw (if staffing allows). Next, participants will be given 90 minutes to use ad lib, i.e., as much as desired.
  Interventions: Other: Subox Mini C with Avail 18 mg nicotine salt (protonated); Other: Subox Mini C with Avail 18 mg nicotine (unprotonated); Other: Own brand cigarette
- ENDS with protonated nicotine first, then Own brand cigarette, then ENDS with unprotonated nicotine (Experimental): In each of the 3 sessions, participants will be instructed to take one puff of the tobacco product (cigarette or Subox Mini C ENDS with 18 mg nicotine) every 30 seconds for 5 minutes followed by a 2nd blood draw (if staffing allows). Next, participants will be given 90 minutes to use ad lib, i.e., as much as desired.
  Interventions: Other: Subox Mini C with Avail 18 mg nicotine salt (protonated); Other: Subox Mini C with Avail 18 mg nicotine (unprotonated); Other: Own brand cigarette
- ENDS with protonated nicotine first, then ENDS with unprotonated nicotine, then Own brand cigarette (Experimental): In each of the 3 sessions, participants will be instructed to take one puff of the tobacco product (cigarette or Subox Mini C ENDS with 18 mg nicotine) every 30 seconds for 5 minutes followed by a 2nd blood draw (if staffing allows). Next, participants will be given 90 minutes to use ad lib, i.e., as much as desired.
  Interventions: Other: Subox Mini C with Avail 18 mg nicotine salt (protonated); Other: Subox Mini C with Avail 18 mg nicotine (unprotonated); Other: Own brand cigarette
- Own brand cigarette first, then ENDS with unprotonated nicotine, then ENDS with protonated nicotine (Experimental): In each of the 3 sessions, participants will be instructed to take one puff of the tobacco product (cigarette or Subox Mini C ENDS with 18 mg nicotine) every 30 seconds for 5 minutes followed by a 2nd blood draw (if staffing allows). Next, participants will be given 90 minutes to use ad lib, i.e., as much as desired.
  Interventions: Other: Subox Mini C with Avail 18 mg nicotine salt (protonated); Other: Subox Mini C with Avail 18 mg nicotine (unprotonated); Other: Own brand cigarette
- ENDS with unprotonated nicotine first, then Own brand cigarette, then ENDS with protonated nicotine (Experimental): In each of the 3 sessions, participants will be instructed to take one puff of the tobacco product (cigarette or Subox Mini C ENDS with 18 mg nicotine) every 30 seconds for 5 minutes followed by a 2nd blood draw (if staffing allows). Next, participants will be given 90 minutes to use ad lib, i.e., as much as desired.
  Interventions: Other: Subox Mini C with Avail 18 mg nicotine salt (protonated); Other: Subox Mini C with Avail 18 mg nicotine (unprotonated); Other: Own brand cigarette

INTERVENTIONS:
Other: Subox Mini C with Avail 18 mg nicotine salt (protonated) — Participants will be instructed to take one puff of the Subox Mini C with Avail 18 mg nicotine salt (protonated) liquid every 30 seconds for 5 minutes followed by a 2nd blood draw. Next, participants will be given 90 minutes to use the product ad lib, i.e., as much as desired.
Other: Subox Mini C with Avail 18 mg nicotine (unprotonated) — Participants will be instructed to take one puff of the Subox Mini C with Avail 18 mg nicotine (unprotonated) liquid every 30 seconds for 5 minutes followed by a 2nd blood draw. Next, participants will be given 90 minutes to use the product ad lib, i.e., as much as desired.
Other: Own brand cigarette — Participants will be instructed to take one puff of a cigarette matching their typical brand every 30 seconds for 5 minutes followed by a 2nd blood draw. Next, participants will be given 90 minutes to use the product ad lib, i.e., as much as desired.

SUMMARY:
This grant compares the effects of cigarette smoking, protonated nicotine ("salt") aerosol through an Electronic Nicotine Delivery System (ENDS), and unprotonated nicotine aerosol through an ENDS on nicotine delivery, nicotine craving, and other outcomes in cigarette smokers.

DETAILED DESCRIPTION:
The purpose of this study is to determine differences in nicotine delivery, user behavior, subjective effects, and physiological effects, when cigarette smokers use a nicotine "salt" (protonated) aerosol, relative to an unprotonated aerosol or their own brand of cigarettes.

ELIGIBILITY:
Inclusion Criteria:

Participants must be:

* healthy (determined by self-report)
* between 21-55 years old
* wiling to provide informed consent
* able to attend lab and abstain from tobacco/nicotine as required and agree to use designated products according to study protocol
* cigarette smokers

Exclusion Criteria:

• Women if breast-feeding or test positive for pregnancy (by urinalysis) at screening

Some study details about eligibility criteria are purposely omitted at this time to preserve scientific integrity. Full details will be posted at the conclusion of the study.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul T Harrell, Ph.D., Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a within-subjects design study with 3 conditions on 3 separate follow-ups after an initial screening visit. Enrolled participants were sometimes excluded from the study, primarily due to loss to follow-up.
Period: Overall Study
Arm/Group | Own Brand Cigarette First, Then ENDS With Protonated Nicotine, Then ENDS With Unprotonated Nicotine | ENDS With Unprotonated Nicotine First, Then ENDS With Protonated Nicotine, Then Own Brand Cigarette | ENDS With Protonated Nicotine First, Then Own Brand Cigarette, Then ENDS With Unprotonated Nicotine | ENDS With Protonated Nicotine First, Then ENDS With Unprotonated Nicotine, Then Own Brand Cigarette | Own Brand Cigarette First, Then ENDS With Unprotonated Nicotine, Then ENDS With Protonated Nicotine | ENDS With Unprotonated Nicotine First, Then Own Brand Cigarette, Then ENDS With Protonated Nicotine
Started | 1 | 3 | 1 | 1 | 1 | 4
Completed | 1 | 1 | 1 | 1 | 1 | 0
Not Completed | 0 | 2 | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Study ended early due to COVID and funding delays.
Groups:
- Total: Total of all reporting groups
Arm/Group | Own Brand Cigarette First, Then ENDS With Protonated Nicotine, Then ENDS With Unprotonated Nicotine | ENDS With Unprotonated Nicotine First, Then ENDS With Protonated Nicotine, Then Own Brand Cigarette | ENDS With Protonated Nicotine First, Then Own Brand Cigarette, Then ENDS With Unprotonated Nicotine | ENDS With Protonated Nicotine First, Then ENDS With Unprotonated Nicotine, Then Own Brand Cigarette | Own Brand Cigarette First, Then ENDS With Unprotonated Nicotine, Then ENDS With Protonated Nicotine | ENDS With Unprotonated Nicotine First, Then Own Brand Cigarette, Then ENDS With Protonated Nicotine | Total
Number analyzed (Participants) | 1 | 3 | 1 | 1 | 1 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (0) | 34.7 (8.5) | 38 (0) | 30 (0) | 41 (0) | 40.8 (10.9) | 34.3 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 0 | 0 | 4 | 7
  Male | 0 | 2 | 0 | 1 | 1 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 3 | 1 | 1 | 1 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 0 | 1 | 1 | 6
  White | 0 | 0 | 1 | 0 | 0 | 2 | 3
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 1 | 1 | 1 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Plasma Nicotine
Description: Change in plasma nicotine level
Time Frame: Blood will be taken 4 times in each session: baseline, 5 minutes after the start of a 10-puff product use, and then before and after an approximately 1-hour ad lib use period.
Population: We were unable to collect this outcome measure (plasma nicotine) due to staffing issues and difficulties with blood draws.
Groups:
- Own Brand Cigarette: Participants will be instructed to take one puff of the tobacco product (cigarette or ENDS) every 30 seconds for 5 minutes followed by a 2nd blood draw. Next, participants will be given 90 minutes to use ad lib, i.e., as much as desired.
  Own brand cigarette: Participants will be instructed to take one puff of a cigarette matching their typical brand every 30 seconds for 5 minutes followed by a 2nd blood draw. Next, participants will be given 90 minutes to use the product ad lib, i.e., as much as desired.
- ENDS: Subox Mini C With 18 mg Nicotine Salt (Protonated): Participants will be instructed to take one puff of the tobacco product (cigarette or ENDS) every 30 seconds for 5 minutes followed by a 2nd blood draw. Next, participants will be given 90 minutes to use ad lib, i.e., as much as desired.
  Subox Mini C with Avail 18 mg nicotine salt (protonated): Participants will be instructed to take one puff of the Subox Mini C with Avail 18 mg nicotine salt (protonated) liquid every 30 seconds for 5 minutes followed by a 2nd blood draw. Next, participants will be given 90 minutes to use the product ad lib, i.e., as much as desired.
- ENDS: Subox Mini C With 18 mg Nicotine Regular (Unprotonated): Participants will be instructed to take one puff of the tobacco product (cigarette or ENDS) every 30 seconds for 5 minutes followed by a 2nd blood draw. Next, participants will be given 90 minutes to use ad lib, i.e., as much as desired.
  Subox Mini C with Avail 18 mg nicotine (unprotonated): Participants will be instructed to take one puff of the Subox Mini C with Avail 18 mg nicotine (unprotonated) liquid every 30 seconds for 5 minutes followed by a 2nd blood draw. Next, participants will be given 90 minutes to use the product ad lib, i.e., as much as desired.
Arm/Group | Own Brand Cigarette | ENDS: Subox Mini C With 18 mg Nicotine Salt (Protonated) | ENDS: Subox Mini C With 18 mg Nicotine Regular (Unprotonated)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Own Brand Cigarette | ENDS: Subox Mini C With 18 mg Nicotine Salt (Protonated) | ENDS: Subox Mini C With 18 mg Nicotine Regular (Unprotonated)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT03974152/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT03974152/ICF_001.pdf